CLINICAL TRIAL: NCT00784654
Title: A Phase III, Double-blind, Placebo-controlled, Randomised Withdrawal, Multicentre, Extension, Safety and Efficacy Study of Lisdexamfetamine Dimesylate (LDX) in Children and Adolescents Aged 6-17 With Attention- Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Double-blind, Placebo-controlled, Randomised Withdrawal, Extension, Safety and Efficacy Study of LDX in Children and Adolescents Aged 6-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-326; 2008-000720-10 (EudraCT Number)
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Lisdexamfetamine dimesylate (LDX) (Experimental): Open-label 30, 50, or 70mg
  Interventions: Drug: Lisdexamfetamine dimesylate (LDX)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate (LDX) — LDX 30, 50, or 70mg capsule once per day (open-label and double-blind periods)
  Other Names: Vyvanse, SPD489
  Arms: Lisdexamfetamine dimesylate (LDX)
Drug: Placebo — Placebo capsule once per day (double-blind period)
  Arms: Placebo

SUMMARY:
The main aim of this study is to evaluate the long-term maintenance of efficacy of LDX after administered to children and adolescents aged 6-17 with ADHD for at least 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent or legally authorised representative(LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations before completing any study-related procedures.
2. Subject and parent/LAR are willing and able to comply with all the testing and requirements defined in this protocol, including oversight of morning dosing. Specifically, the parent/LAR must be available upon awakening, at approximately 7:00AM, to dispense the dose of test product for the duration of the study.
3. Subject is a male or female aged 6-17 years inclusive at the time of consent for the antecedent study (SPD489-325).
4. Subject satisfied all entry criteria for the antecedent study (SPD489-325), and completed a minimum of 4 weeks of double-blind treatment, reached Visit 4 and completed the 1-week post-treatment washout in the antecedent study (SPD489-325), without experiencing any clinically significant AEs that would preclude exposure to LDX.
5. Subject must have a satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination findings and clinical laboratory test results.
6. Subject has blood pressure measurements within the 95th percentile for age, gender, and height.

Exclusion Criteria:

1. Subject was terminated from SPD489-325 for non-compliance and/or experienced an SAE or AE resulting in termination from the antecedent study.
2. Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any severe comorbid Axis II disorder or severe Axis I disorder (such as Post Traumatic Stress Disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder) or other symptomatic manifestations, such as agitated states, marked anxiety, or tension that, in the opinion of the examining clinician, will contraindicate treatment with LDX or confound efficacy or safety assessments. Comorbid psychiatric diagnoses will be established at the Screening Visit (Visit -1)of the antecedent study (SPD489-325)with the Screening interview of the Kiddie-SADS-Present and Lifetime-Diagnostic Interview (K-SADS-PL)and additional modules if warranted by the results of the initial interview. Participation in behavioural therapy is permitted provided the subject was receiving the therapy for at least 1 month at the time of the Baseline Visit (Visit 0) of the antecedent study (SPD489-325).
3. Subject has a conduct disorder. Oppositional defiant disorder is not exclusionary.
4. Subject has any concurrent chronic or acute illness or unstable medical condition that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
5. Subject is currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently, demonstrating active suicidal ideation.
6. Subject is female and is pregnant or lactating.
7. Subject has glaucoma.
8. Subject has any clinically significant ECG at Visit 8 of the antecedent study (SPD489-325) or clinically significant laboratory abnormalities at Visit 7 of the antecedent study (SPD489-325).
9. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine.
10. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine)in accordance with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR)criteria.
11. Subject has a history of seizures (other than infantile febrile seizures), a tic disorder, a current diagnosis and or a known family history of Tourette's Disorder.
12. Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
13. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
14. Subject is taking any medication that is excluded.
15. Subject is taking other medications that have central nervous system (CNS) effects, affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors (during or within 14 days of investigational medicinal product administration). Stable use of bronchodilator inhalers is not exclusionary.
16. Subject has a documented allergy, hypersensitivity, or intolerance to any excipients in the investigational medicinal product(s).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2009-01-27 (Actual); Primary Completion 2011-10-26 (Actual); Study Completion 2011-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (51):
- United States (4):
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Miami Research Associates, South Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - CNS Healthcare, Memphis, Tennessee
- Belgium (3):
  - ZNA Antwerpen, Commandant Weynsstraat 165, Hoboken, Antwerpen
  - Afdeling Psychiatrie, UZ Herestraat 49, Leuven, Flemish Brabant
  - Universitair Ziekenhuis Gent, Kinder - en Jeugdpsychiatrie, Ghent, Oost-vlaanderen
- France (3):
  - Hôpital Gui de Chauliac, Montpellier
  - Hospital Archet 2, Nice
  - Hôpital Robert Debré, Paris, Île-de-France Region
- Germany (15):
  - Albert-Ludwigs-Universitat Freiburg, Freiburg im Breisgau, Baden-wuttemberg
  - Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim, Baden-wuttemberg
  - Schwerpunktpraxis für Entwicklung und Lernen, Bamberg, Bavaria
  - Medizinisches Studienzentrum Würzburg, Würzburg, Bavaria
  - Universität Würzburg, Würzburg, Bavaria
  - Institutsambulanz Bad Nauheim, Bad Nauheim, Hesse
  - Universitat Göttingen, Göttingen, Lower Saxony
  - Universität zu Köln, Klinik und Poliklinik für Psychiatrie und Psychotherapie des Kindes und Jugendalters, Cologne, North Rhine-Westphalia
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsmedizin Berlin, Berlin
  - Praxis Dr. Walter Robert Otto, Fulda
  - Praxis Dr. Wolff, Hagen
  - Praxis für Neuropädiatrie, Hamburg
  - Praxis Dr med. Friedrich Kaiser und Dr. med. Ingrid Marinesse, Hamburg
  - Universitätsklinikum Gießen und Marburg GmbH, Universitätsklinikum Gießen und Marburg GmbH, Hans-Sachs-Straße 4,, Marburg
- Hungary (4):
  - Vadaskert Kórház és Szakambulancia, Budapest
  - Pándy Kálmán Kórház, Gyula
  - Gyermek és Ifjúságpszichiátriai Szakrendelés és Gondozó, Pécs
  - Szegedi Tudományegyetem, Szeged
- Italy (4):
  - Azienda Ospedaliera Policlinico Consorziale, Bari
  - Università degli Studi di Cagliari, Cagliari
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Azienda Ospedaliera della 2? Universita di Napoli, Napoli
- Poland (5):
  - Specjalistyczna Praktyka Lekarska, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki im. dr. Antoniego Jurasza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewódzki Osrodek Lecznictwa Psychiatrycznego, Torun, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Poradnia Psychiatryczna, ul. Marszalkowska 24,, Warsaw, Masovian Voivodeship
  - Gdanski Uniwersytet Medyczna w Gdansku, Gdansk, Pomeranian Voivodeship
- Sweden (4):
  - Drottning Silvias Barnsjukhus, Otterhällegatan 12A, Gothenburg
  - Utvecklingsneurologiska Enheten (UNE), Mariestad
  - Astrid Lindgren Children's Hospital, Karolinska University Hospital, Stockholm
  - Barn och Ungdomsmedicin klinik Mölnlycke, Stockholm
- United Kingdom (9):
  - Parkview Clinic, Birmingham, England
  - East Kent NHS and Social Care Partnership Trust, Ramsgate, England
  - Lighthouse Child Development Centre, Southend-on-Sea, Essex
  - Victoria Hospital, Paediatric Unit, Kirkcaldy, FIFE
  - Tayside Children's Hospital, Dundee, Scotland
  - Ryegate Children's Centre, Sheffield, Yorkshire
  - Basildon Hospital - Child Development Centre,, Basildon
  - Northampton Child and Adolescent Mental Health Services, Northampton
  - Child and Family Mental Health Services, Wigan

REFERENCES:
- [Derived] Banaschewski T, Johnson M, Lecendreux M, Zuddas A, Adeyi B, Hodgkins P, Squires LA, Coghill DR. Health-related quality of life and functional outcomes from a randomized-withdrawal study of long-term lisdexamfetamine dimesylate treatment in children and adolescents with attention-deficit/hyperactivity disorder. CNS Drugs. 2014 Dec;28(12):1191-203. doi: 10.1007/s40263-014-0193-z. PMID 25139785
- [Derived] Coghill DR, Banaschewski T, Lecendreux M, Johnson M, Zuddas A, Anderson CS, Civil R, Dauphin M, Higgins N, Lyne A, Gasior M, Squires LA. Maintenance of efficacy of lisdexamfetamine dimesylate in children and adolescents with attention-deficit/hyperactivity disorder: randomized-withdrawal study design. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):647-657.e1. doi: 10.1016/j.jaac.2014.01.017. Epub 2014 Mar 4. PMID 24839883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Open-label period, 8 subjects completed the Open-label period and were not randomized. Therefore, 157 subjects were randomized in the Randomized Withdrawal Period.
Groups:
- Lisdexamfetamine Dimesylate (LDX)(Open-label Period): Consists of at least 26 weeks where subjects are titrated to an optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours) and then maintained on their optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours).
- Lisdexamfetamine Dimesylate (LDX)(Randomized Period): After the Open-label Period, subjects were randomized to receive their optimal dose of LDX at either 30, 50, or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours for up to 6 weeks.
- Placebo (Randomized Period): After the Open-label Period, subjects were randomized to receive placebo once-daily orally at approximately 7:00 AM +/- 2 hours for up to 6 weeks.
Period: Open-Label Period (Non-Randomized)
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period) | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Started | 276 | 0 | 0
Completed | 165 | 0 | 0
Not Completed | 111 | 0 | 0
Not completed — Adverse Event | 44 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 0 | 0
Not completed — Lack of Efficacy | 21 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0
Not completed — Mother is a drug addict | 1 | 0 | 0
Not completed — Decision of medical monitor | 1 | 0 | 0
Not completed — Home situation intolerable | 1 | 0 | 0
Not completed — ADHD-RS score too high for Random Phase | 1 | 0 | 0
Not completed — Met stopping criteria for CGI-S score | 1 | 0 | 0
Not completed — Did not provide end of study page | 1 | 0 | 0
Period: Randomized Withdrawal Period
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period) | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Started | 0 | 78 | 79
Completed | 0 | 60 | 16
Not Completed | 0 | 18 | 63
Not completed — Met relapse criteria per investigator | 0 | 8 | 35
Not completed — Lack of Efficacy | 0 | 5 | 18
Not completed — Withdrawal by Subject | 0 | 1 | 7
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Did not complete a visit | 0 | 1 | 0
Not completed — Family reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (2.82)
Age, Customized [Count of Participants; unit: Participants]
  6-12 years | 191
  13-17 years | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 212
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
  Italy | 20
  United Kingdom | 16
  France | 11
  Hungary | 28
  Belgium | 9
  Poland | 8
  Germany | 95
  Sweden | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Treatment Failures at End of The Randomized Withdrawal Period
Description: Treatment failure defined as 50% increase (worsening) in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) total score and >= 2 point increase (worsening) in the Clinical Global Impression-Severity of Illness (CGI-S) score observed at any visit during the randomized withdrawal period compared to the respective scores at baseline of randomized withdrawal period. Subjects without an endpoint value were classed as treatment failures.
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized Full Analysis Set (Randomized FAS) includes all subjects who were randomized and received at least 1 dose of investigational product during the Randomized Withdrawal Period.
Measure: Number; unit: percentage of participants
Groups:
- Lisdexamfetamine Dimesylate (LDX)(Randomized Period): Subjects receive their optimal dose of LDX at either 30, 50, or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours for 6 weeks.
- Placebo (Randomized Period): Subjects receive placebo once-daily orally at approximately 7:00 AM +/- 2 hours for 6 weeks.
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 76 | 77
percentage of participants | 15.8 | 67.5
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Change From Open-Label Baseline in The Attention Deficit Hyperactivity Disorder Rating Scale-Fourth Edition (ADHD-RS-IV) Total Score at Endpoint (Week-26) of The Open-label Period
Description: ADHD-RS-IV consists of 18 items scored on a 4-point scale from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. A decrease in score indicates an improvement in ADHD symptomology.
Time Frame: Open-label baseline and Endpoint (Week-26)
Population: Open-label Full Analysis set (Open-label FAS) includes all subjects who received at least 1 dose of investigational product during the Open-label Period.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 257
Scores on a scale | -26.6 (11.39)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Open-label Period); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Randomized Withdrawal Baseline in The ADHD-RS-IV Total Score at Endpoint of The Randomized Withdrawal Period
Description: as for outcome 2
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Lisdexamfetamine Dimesylate (LDX)(Randomized Period): Subjects receive their optimal dose of LDX at either 30, 50, or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours for up to 6 weeks.
- Placebo (Randomized Period): Subjects receive placebo once-daily orally at approximately 7:00 AM +/- 2 hours for up to 6 weeks.
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 73 | 73
Scores on a scale | 1.2 (1.09) | 13.8 (1.06)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-15.4 to -9.8]

4. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Endpoint (Week-26) of The Open-label Period
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: At Week 26
Population: Open-label FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 198
percentage of participants
  Normal, not at all ill | 39.9
  Borderline mentally ill | 46.5
  Mildly ill | 1.5
  Moderately ill | 6.6
  Markedly ill | 4.5
  Severely ill | 0.5
  Among the most extremely ill | 0.5

5. Other Pre Specified Outcome: Percent of Participants With CGI-S at Open-label Baseline
Description: as for outcome 4
Time Frame: Open-label baseline
Population: Open-label FAS
Measure: Number; unit: percentage of participants
Groups:
- Lisdexamfetamine Dimesylate (LDX)(Open-label Period): Consists of at least 26 weeks where subjects are titrated to an optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours) and then maintained on their optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM +/- 2 hours ).
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 261
percentage of participants
  Normal, not at all ill | 0
  Borderline mentally ill | 0
  Mildly ill | 1.5
  Moderately ill | 27.2
  Markedly ill | 50.2
  Severely ill | 17.6
  Among the most extremely ill | 3.4

6. Secondary Outcome: Percent of Participants With CGI-S at Endpoint of The Randomized Withdrawal Period, Last Observation Carried Forward (LOCF)
Description: as for outcome 4
Time Frame: At endpoint of the randomized withdrawal period (Up to 6 weeks)
Population: Randomized FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 75 | 73
percentage of participants
  Normal, not at all ill | 40.0 | 8.2
  Borderline mentally ill | 41.3 | 19.2
  Mildly ill | 8.0 | 11.0
  Moderately ill | 10.7 | 39.7
  Markedly ill | 0 | 15.1
  Severely ill | 0 | 6.8
  Among the most extremely ill | 0 | 0
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percent of Participants With Improvement on Clinical Global Impression - Improvement (CGI-I) at Endpoint (Week-26) of The Open-label Period
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale. Improvement includes CGI-I categories of very much improved and much improved. No improvement includes all other assessed categories.
Time Frame: At Week 26
Population: Open-label FAS
Measure: Number; unit: percentage of improved participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 257
percentage of improved participants | 79.8

8. Secondary Outcome: Change From Open-label Baseline in The Health Utilities Index-2 (HUI-2) Scores at Endpoint (Week-26) of The Open-label Period, LOCF
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status.
Time Frame: At open-label baseline and endpoint (Week-26) of the open-label period
Population: Open-label FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 223
scores on a scale | 0.087 (0.1307)

9. Secondary Outcome: Change From Randomized Withdrawal Baseline in The HUI-2 Scores at Endpoint of The Randomized Withdrawal Period
Description: as for outcome 8
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 59 | 62
Scores on a scale | -0.005 (0.0772) | -0.046 (0.1098)

10. Secondary Outcome: Change From Open-label Baseline in The Child Health and Illness Profile, Child Edition: Parent Report Form (CHIP-CE:PRF) Global T-score at Endpoint (Week-26) of The Open-label Period
Description: The CHIP-CE:PRF evaluates health-related quality of life. It is composed of 5 domains (satisfaction, comfort, resilience, avoidance, and achievement) consisting of a total of 76 items. The global score is an average of the scores for the 5 domains. The majority of items assess frequency of events using a 5-point response format. There is no range for a total score. Raw scale scores are used to generate T-scores. Higher scores indicate better health.
Time Frame: At open-label baseline and endpoint (Week-26) of the open-label period
Population: Open-label FAS
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 207
T-scores | 10.2 (10.71)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Open-label Period); Test type: Superiority or Other; p < 0.001, t-test, 1 sided

11. Secondary Outcome: Change From Randomized Withdrawal Baseline in The CHIP-CE:PRF Global T-score at Endpoint of The Randomized Withdrawal Period
Description: as for outcome 10
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 52 | 60
T-scores | 1.1 (1.17) | -5.4 (1.10)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [3.5 to 9.5]

12. Secondary Outcome: Change From Open-Label Baseline in The Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Global Score at Endpoint (Week-26) of The Open-label Period
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: At open-label baseline and endpoint (Week-26) of the open-label period
Population: Open-label FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 223
scores on a scale | -0.43 (0.42)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Open-label Period); Test type: Superiority or Other; p < 0.001, t-test, 1 sided

13. Secondary Outcome: Change From Randomized Withdrawal Baseline in The WFIRS-P Global Score at Endpoint of The Randomized Withdrawal Period
Description: as for outcome 12
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 58 | 61
Scores on a scale | 0.01 (0.03) | 0.20 (0.03)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.26 to -0.11]

14. Secondary Outcome: Change From Open-Label Baseline in The Brief Psychiatric Rating Scale for Children (BPRS-C) Total Score at Endpoint (Week-26) of The Open-label Period
Description: The BPRS-C characterizes psychopathology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology.
Time Frame: At open-label baseline and endpoint (Week-26) of the open-label period
Population: Open-label Safety Population includes all subjects who received at least 1 dose of investigational product in the Open-label period.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 84
Scores on a scale | -13.9 (12.58)

15. Secondary Outcome: Change From Randomized Withdrawal Baseline in BPRS-C Total Score at Endpoint of The Randomized Withdrawal Period
Description: as for outcome 14
Time Frame: Baseline of the randomized withdrawal period and its relevant endpoint (Up to 6 weeks)
Population: Randomized Safety Population includes all subjects who received at least 1 dose of any investigational product during the Randomized Withdrawal Period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 23 | 27
Scores on a scale | -17.1 (11.17) | -9.1 (11.26)

16. Other Pre Specified Outcome: Percent of Participants With CGI-S at Randomized Withdrawal Baseline
Description: as for outcome 4
Time Frame: Randomized withdrawal baseline
Population: Randomized FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 74 | 77
percentage of participants
  Normal, not at all ill | 50.0 | 46.8
  Borderline mentally ill | 50.0 | 53.2
  Mildly ill | 0 | 0
  Moderately ill | 0 | 0
  Markedly ill | 0 | 0
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX)(Randomized Period) vs Placebo (Randomized Period); Test type: Superiority or Other; p = 0.726, Cochran-Mantel-Haenszel

17. Other Pre Specified Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) During The Open-label Period
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: From open-label baseline to Week-26
Population: Open-label Safety Population
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period)
Number analyzed (Participants) | 118
participants
  Suicidal ideation | 1
  Suicidal behavior | 0

18. Other Pre Specified Outcome: C-SSRS During the Randomized Withdrawal Period
Description: as for outcome 17
Time Frame: Baseline of the randomized withdrawal period to end of the study (Up to 6 weeks)
Population: Randomized Safety Population
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Number analyzed (Participants) | 45 | 41
participants
  Suicidal ideation | 0 | 0
  Suicidal behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: 33 weeks
Groups:
- Lisdexamfetamine Dimesylate (LDX)(Open-label Period): Consists of at least 26 weeks where subjects are titrated to an optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM) and then maintained on their optimal dose of LDX (either 30, 50 or 70 mg once-daily orally at approximately 7:00 AM).
- Lisdexamfetamine Dimesylate (LDX)(Randomized Period): After the Open-label Period, subjects were randomized to receive their optimal dose of LDX at either 30, 50, or 70 mg once-daily orally at approximately 7:00 AM for up to 6 weeks.
- Placebo (Randomized Period): After the Open-label Period, subjects were randomized to receive placebo once-daily orally at approximately 7:00 AM for up to 6 weeks.
Arm/Group | Lisdexamfetamine Dimesylate (LDX)(Open-label Period) | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) | Placebo (Randomized Period)
Serious Adverse Events (participants affected / at risk) | 12/276 | 0/78 | 1/79
Other Adverse Events (participants affected / at risk) | 227/276 | 31/78 | 20/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (LDX)(Open-label Period) (N=276) | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) (N=78) | Placebo (Randomized Period) (N=79)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Treatment noncompliance (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (LDX)(Open-label Period) (N=276) | Lisdexamfetamine Dimesylate (LDX)(Randomized Period) (N=78) | Placebo (Randomized Period) (N=79)
Decreased appetite (Metabolism and nutrition disorders) | 76 (91) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 58 (80) | 6 (6) | 5 (7)
Weight decreased (Investigations) | 46 (60) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 43 (64) | 7 (7) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 41 (48) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 39 (44) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 32 (43) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (36) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 23 (25) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 20 (25) | 2 (2) | 0 (0)
Initial insomnia (Psychiatric disorders) | 20 (22) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 2 (2) | 0 (0)
Fatigue (General disorders) | 18 (22) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 18 (25) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 14 (21) | 1 (1) | 1 (1)
Irritability (General disorders) | 13 (17) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 11 (16) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (9) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (11) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 8 (11) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 7 (7) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 7 (7) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 6 (6) | 1 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.